CLINICAL TRIAL: NCT03229798
Title: An Open-Label Phase 1 Study to Establish the Pharmacokinetics and Safety of Sumatriptan Succinate Administered Via the Sofusa™ DoseConnect™ System at Escalating Doses Compared to Oral Imitrex® Single 100 mg Dose in Healthy Subjects
Brief Title: Sofusa System With Sumatriptan (KC5010) Phase 1 Dose Escalation Safety and PK Study (KCC-SMT-002)
Acronym: KCC-SMT-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Collaborators: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: REC-0000330, Ver 1
Record Dates: First submitted 2017-07-20; First posted 2017-07-26 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Sumatriptan Succinate Oral Tablet (Active Comparator): 100 mg oral tablet commercial Imitrex sumatriptan succinate tablet
  Interventions: Drug: Sumatriptan Succinate Oral Tablet
- Sofusa Profile #1 (Experimental): Combination device for transdermal delivery of sumatriptan succinate Current approved dose (SC)
  Interventions: Combination Product: Transdermal delivery of sumatriptan succinate
- Sofusa Dose Profile #2 (Experimental): Combination device for transdermal delivery of sumatriptan succinate- adjust dose and flow rate to achieve PK profile based on results from Sofusa Dose Profile #1
  Interventions: Combination Product: Transdermal delivery of sumatriptan succinate
- Sofusa Dose Profile #3 (Experimental): Combination device for transdermal delivery of sumatriptan succinate- adjust dose and flow rate to achieve PK profile based on results from Sofusa Dose Profile #2
  Interventions: Combination Product: Transdermal delivery of sumatriptan succinate
- Sofusa Dose Profile #4 (Experimental): Combination device for transdermal delivery of sumatriptan succinate- adjust dose and flow rate to achieve PK profile based on results from Sofusa Dose Profile #3
  Interventions: Combination Product: Transdermal delivery of sumatriptan succinate
- Sofusa Dose Profile #5 (Experimental): Combination device for transdermal delivery of sumatriptan succinate- adjust dose and flow rate to achieve PK profile based on results from prior Sofusa Dose Profile #2-4
  Interventions: Combination Product: Transdermal delivery of sumatriptan succinate

INTERVENTIONS:
Drug: Sumatriptan Succinate Oral Tablet — Sumatriptan succinate commercial Imitrex 100 mg tablet
  Arms: Sumatriptan Succinate Oral Tablet
Combination Product: Transdermal delivery of sumatriptan succinate — Sumatriptan succinate transdermal drug delivery system
  Other Names: Sofusa DoseDisc; Sofusa DoseConnect; KC5010
  Arms: Sofusa Dose Profile #2; Sofusa Dose Profile #3; Sofusa Dose Profile #4; Sofusa Dose Profile #5; Sofusa Profile #1

SUMMARY:
Study KCC-SMT-002, is a Phase 1, single-site, open-label, non-randomized, crossover, flexible dose design study to investigate the pharmacokinetic (PK) and safety comparing the Sofusa™ system with sumatriptan (KC5010) to Imitrex® oral tablets in 17 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give voluntary written informed consent (personally signed and dated) and HIPPA Authorization prior to any study related procedures.
2. Available to participate for the entire study period.
3. Be a male or female person between 18 and 55 years (inclusive) of age.
4. Healthy as determined by the investigator based on a medical evaluation including history, physical examination, electrocardiogram (ECG), and laboratory tests.
5. Have systolic blood pressure (sitting) of < 140 mmHg and diastolic blood pressure of < 90 mmHg after 5 minutes of rest. Minor excursions in blood pressure outside of this range may be acceptable if determined not to be clinically significant by the study physician or medical monitor.
6. Have resting pulse rate (sitting) within normal range of 60-100 bpm. Minor excursions in resting pulse outside of this range may be acceptable if determined not to be clinically significant by the study physician or the medical monitor.
7. Females must be either postmenopausal for at least 1 year, surgically sterile (bilateral oophorectomy, tubal ligation, tubal occlusion, hysterectomy), or using adequate contraception from screening until 90 days after completion of study participation. Adequate contraception is defined as true abstinence, a vasectomized partner, or one of the following in combination with a diaphragm, cervical cap, or a condom:

   * Hormonal contraceptives (oral, implant, patch, injection)
   * Intrauterine device

   Males must use adequate contraception and must not donate sperm from first admission to the clinical research center until 90 days after completion of study participation. Adequate contraception is defined as true abstinence, vasectomy, a partner who is surgically sterile (bilateral oophorectomy, tubal ligation, tubal occlusion, hysterectomy), or one of the following in combination with a diaphragm, cervical cap, or a condom:
   * Hormonal contraceptives (oral, implant, patch, injection)
   * Intrauterine device
8. Have a body weight above 50 kg and below 90 kg (inclusive).
9. Be able to communicate effectively with the study personnel and understand and comply with all study requirements.

Exclusion criteria:

1. Women who are pregnant or lactating.
2. Current use or has used tobacco- or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, etc.) 30 days prior to investigational product administration. A cotinine test (with a cut-off of 200 mg) will be performed at screening and admission to the study center.
3. Recent history (i.e. within 2 years) of alcohol abuse, illicit drug use, or significant mental illness.
4. Positive screen for substances of abuse.
5. A positive screening result for human immunodeficiency virus (HIV) antibody, Hepatitis B surface antigen (HBsAg), or Hepatitis C antibody (anti-HCV).
6. Any disease or condition (medical or surgical) that might compromise a major body system (e.g. cardiovascular, respiratory, etc.) or conditions that may interfere with the absorption, distribution, metabolism, or excretion of the study medication.
7. Any bleeding disorders or use of anticoagulants.
8. Any conditions (e.g. diabetes, edema, scleroderma) or receiving medications (e.g. steroids, antibiotics) that alter skin integrity and/or healing. Any known condition or receiving medications causing hypo/hyperpigmentation or photosensitivity.
9. Presence or history of hypertension or other cardiovascular abnormalities such as, but not limited to, myocardial infarction, heart failure, arrhythmia, stroke, or peripheral vascular disease or any other cardiovascular disease that requires the subject to wear a pacemaker.
10. Use of a drug therapy known to induce or inhibit hepatic drug metabolism within 30 days prior to the Treatment visit for dosing.
11. Patient has received a live attenuated vaccine within the 4 weeks prior to treatment or plans to receive one during the study.
12. Febrile illness within 7 days of Treatment visit for dosing.
13. Has a positive history or known sensitivity to sumatriptan or other triptans.
14. Any history of sensitivity to methylene blue, fluorescein or calcein, or other similar dye product.
15. Subjects who have used ergotamine-containing or ergot-type medications (like dihydrogergotamine or methysergide) within the past week. The Imitrex® label specifies that these medication are contraindicated within 24 hours of use.
16. Diagnosed with ischemic bowel disease or severe hepatic impairment which are known contraindications to sumatriptan.
17. Concomitant therapy with the following medications which have significant drug interactions with sumatriptan: selective serotonin reuptake inhibitors (SSRIs), serotonin/norepinephrine reuptake inhibitor (SNRIs), tricyclic antidepressants, and monomine oxidase (MAO) inhibitors due to an increased risk of serotonin syndrome. Subjects receiving these medications may enroll in the study if these medications have been discontinued for 5 or more half-lives prior to the first Treatment visit.
18. Subjects who are currently taking prescription or over-the-counter medications (including vitamins and herbal preparations) that could interfere with the evaluation or the safety of the subject, as determined by the Investigator.
19. Participation in the treatment phase of a clinical study or receipt of an investigational drug or medical device within 30 days prior to the Treatment visit for dosing.
20. History of difficulty with phlebotomy procedures.
21. Donated blood (>400 mL) or blood products within 45 days prior to the Treatment visit for dosing.
22. Subjects who have skin conditions or tattoos extensive enough to cover areas where the device is to be applied.
23. Any history of skin contact sensitivity to metals, plastics or adhesives.
24. Has a condition that, in the opinion of the Investigator, may increase the risk to the subject and/or the interpretation of the data.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
PK Cmax | 48 hours after dosing begins
  Pharmacokinetic profile with Cmax (maximum concentration) of drug in blood, ng/mL
PK AUC | 48 hours after dosing begins
  Pharmacokinetic profile AUC (area under the curve) of drug in blood, ng-hr/mL

SECONDARY OUTCOMES:
Dermatological skin response (Draize scale) | From Predose to 168 hours after device application
  Skin response as measured on modified Draize scale (erythema, edema, etc.)
Pain of application and wear (VAS scale) | Upon application and after wear
  Pain as reported on Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Wayne L Harper, MD, Principal Investigator — Carolina Phase I Research, LLC
Locations (1):
- Carolina Phase 1 Research, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kam KR, Walsh LA, Bock SM, Koval M, Fischer KE, Ross RF, Desai TA. Nanostructure-mediated transport of biologics across epithelial tissue: enhancing permeability via nanotopography. Nano Lett. 2013 Jan 9;13(1):164-71. doi: 10.1021/nl3037799. Epub 2012 Dec 24. PMID 23186530
- [Background] Walsh L, Ryu J, Bock S, Koval M, Mauro T, Ross R, Desai T. Nanotopography facilitates in vivo transdermal delivery of high molecular weight therapeutics through an integrin-dependent mechanism. Nano Lett. 2015 Apr 8;15(4):2434-41. doi: 10.1021/nl504829f. Epub 2015 Mar 27. PMID 25790174
- [Background] Owen K, Hartley K, Tucker ML, Parkinson MM, Tweats DJ, Jackson MR. The preclinical toxicological evaluation of sumatriptan. Hum Exp Toxicol. 1995 Dec;14(12):959-73. doi: 10.1177/096032719501401205. PMID 8962747
- See also: Imitrex® oral prescribing information (November 2013) — https://www.gsksource.com/pharma/content/dam/GlaxoSmithKline/US/en/Prescribing_Information/Imitrex_Tablets/pdf/IMITREX-TABLETS-PI-PIL.PDF